CLINICAL TRIAL: NCT04387058
Title: Incidence of Diabetes and Metabolic Disorders After TIPS in Cirrhotic Patients
Acronym: Gluco-TIPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: RC31/18/0361
Record Dates: First submitted 2020-05-09; First posted 2020-05-13 (Actual); Last update posted 2020-05-13 (Actual); Status verified 2020-05

CONDITIONS: Cirrhosis Portal
MeSH Terms: interventions — Portasystemic Shunt, Transjugular Intrahepatic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- patients with cirrhosis and and portal hypertension (Other): All major patients under 70 years of age with cirrhosis and portal hypertension justifying a treatment with TIPS. These patients must be affiliated to a social security and able to sign a free, informed and written consent.
  Interventions: Device: TIPS

INTERVENTIONS:
Device: TIPS — TIPS (Transjugular Intrahepatic Portosystemic Shunt) is an interventional radiology method that creates an anastomosis between the portal venous network and the hepatic venous network.

SUMMARY:
Decompensated cirrhosis is associated with sarcopenia. TIPS is an efficient treatment of portal hypertension. Based on our retrospective data, TIPS induces in 30% of cirrhotic patients metabolic disorders associated with diabetes or pre-diabetes. The main objective is to measure the cumulative incidence of diabetes and pre-diabetes 6 months after TIPS insertion.

DETAILED DESCRIPTION:
Based on our retrospective data, we expect that one-third of cirrhotic patients develop glucose dysregulation after TIPS. A better knowledge of the metabolic disorders related to the TIPS could allow to prevent the deleterious effects of the TIPS on the disease (decrease of the insulin-sensitivity, fat gain ...), by simple interventions on diet or physical activity. We will assess the incidence of diabetes and pre-diabetes, and the influence of TIPS on nutritional status and sarcopenia. Patients will be follow-up 6 months after TIPS. We will explore the hormonal mechanisms that explain these changes.

ELIGIBILITY:
Inclusion Criteria:

* patient cirrhosis and portal hypertension justifying a treatment with TIPS
* written consent.

Exclusion Criteria:

* contraindication for TIPS
* indications of TIPS in emergency or as part of the preparation for a surgical procedure,
* hepatocellular carcinoma outside Milan criteria or cancer at a palliative stage,
* a contra-indication to the realization of an OGTT,
* a hyperglycemic treatment (corticosteroids, somatostatin, etc.),
* hemoglobin <7 g / dl,
* patients who have had a liver transplant,
* those for whom the follow-up is considered impossible or the vital prognosis is engaged in the short term,
* pregnant or lactating women,
* those unable to receive enlightened information,
* those participating in interventional research
* and finally the persons placed under safeguard of justice, tutelage or curatorship.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 111 (Estimated)
Dates: Start 2019-06-16 (Actual); Primary Completion 2022-06-16 (Estimated); Study Completion 2022-06-16 (Estimated)

PRIMARY OUTCOMES:
the cumulative incidence | 6 months
  The primary outcome is the cumulative incidence (%) of diabetes and pre-diabetes observed 6 months after TIPS insertion (M6). Diabetes and pre-diabetes will be defined according to World Health Organization (WHO) criteria, based on fasting blood glucose level or 2h after an oral glucose test

CONTACTS AND LOCATIONS:
Overall Officials: Maeva GUILLAUME, Principal Investigator — University Hospital, Toulouse
Locations (1):
- CHU de Toulouse, Toulouse, Haute-garonne, France